CLINICAL TRIAL: NCT04738240
Title: A Randomised Feasibility Study Into the Use of Endoscopic Visualisation of Rectal Anastomosis vs. Current Practice and the Effect on Anastomotic Leak Rates in Patients Undergoing Rectal Surgery for Bowel Cancer in a Tertiary Referral Centre
Brief Title: Endoscopic Visualisation of Anastomosis in Colorectal Cancer Surgery
Acronym: EVACCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Benjamin William Peter Rossi, Research Fellow, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18/19-1071; 246332 (Other: IRAS)
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer; Colorectal Cancer; Anastomotic Leak; Intraoperative Endoscopy
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-operative endoscopy (Experimental): The intervention arm will have an intra-operative endoscopy performed per rectum once the anastomosis has been performed. The anastomosis will be graded from 1 to 3 in the endoscopic group. Grade 1 is defined as circumferentially normal appearing peri-anastomotic mucosa. Grade 2 is defined as ischemia or congestion involving <30% of either the colon or rectal mucosa. Grade 3 is defined as ischemia or congestion involving >30% of the colon or rectal mucosa or ischemia/congestion involving both sides of the staple line. If appearances are grade 2 a suture re-inforcement or re-anastomosis will be performed; if appearances are grade 3 a re-anastomosis will be performed. Images will be obtained via the endoscopy stack during the assessment.
  Interventions: Diagnostic Test: Intra-operative endoscopy
- Standard air leak test (No Intervention): The control arm will receive an intra-operative leak test. This involves insufflation of air per rectum via bladder syringe while the anastomosis is bathed in sterile water. The presence of air bubbles from the anastomosis denotes a positive test.

INTERVENTIONS:
Diagnostic Test: Intra-operative endoscopy — Intra-operative endoscopy to assess rectal anastomosis
  Arms: Intra-operative endoscopy

SUMMARY:
A randomised feasibility study into the use of endoscopic visualisation of rectal anastomosis vs. current practice and the effect on anastomotic leak rates in patients undergoing rectal surgery for bowel cancer in a tertiary referral centre

DETAILED DESCRIPTION:
Anastomotic leak is one of the biggest challenges in colorectal surgery with little still known about what causes a leak. An anastomotic leak is defined as a defect of the intestinal wall at the anastomotic site leading to a communication between the intra- and extra-luminal compartments. Current leak rates following rectal surgery are between 8% and 17%, which is significant given the numbers of resections performed in our unit, approximately 750 per year. The morbidity of an anastomotic leak can be significant. Most require re-operation and those that do not may require interventional radiological drainage or prolonged hospital stay for intra-venous antibiotics. There is also a high risk of mortality, especially for those requiring a further operation where it can be up to 5.8%. The cost of a leak has been shown to be significant both in monetary terms and by increasing the length of stay. In a study from the USA per 1,000 patients undergoing colorectal surgery, the economic burden associated with anastomotic leaks--including hospitalization and re-admission--was established as 9,500 days in prolonged LOS and $28.6 million in additional costs.

The investigators plan to perform an intra-operative endoscopy for participants undergoing rectal resection and anastomosis to understand what leads to an anastomotic leak and to try and reduce the rates of anastomotic leakage by fixing these problems at the time of operation so they do not lead to a post-operative complication. In the intervention group during the procedure the investigators will visualise the anastomosis endoscopically looking for defects, areas of ischaemia and congestion. Previous retrospective studies have proven the safety of this technique and significant reduction of leak rates, albeit within the limitations of a retrospective study; the investigators plan to take this hypothesis further to using a randomised approach. The anastomosis will be graded from 1 to 3 in the endoscopic group. Grade 1 is defined as circumferentially normal appearing peri-anastomotic mucosa. Grade 2 is defined as ischemia or congestion involving <30% of either the colon or rectal mucosa. Grade 3 is defined as ischemia or congestion involving >30% of the colon or rectal mucosa or ischemia/congestion involving both sides of the staple line. If appearances are grade 2 a suture re-inforcement or re-anastomosis will be performed; if appearances are grade 3 a re-anastomosis will be performed. Images will be taken during the procedure to document the findings.

This compares to current standard practice in the control group of air insufflation into the rectum while the anastomosis is bathed in sterile water to look for the presence of air bubbles which may have come through an anastomotic defect. If the test is positive the surgeon makes a decision regarding whether suture re-inforcement, re-do of the anastomosis and/or defunctioning stoma is required. There are no standardised guidelines for this decision making process. This is currently standard practice in most colorectal departments in the UK.

The aim of the study is to see if this trial design is feasible within the investigators department and if so to progress to a full scale trial. The secondary aim is from the preliminary data to see if there is a significant difference in anastomotic leak rates between participants who receive standard care and participants who receive our intervention. There are no previous randomised trials into this subject and considering the significance of an anastomotic leak we feel this justifies further research.

For patients an anastomotic leak can be catastrophic, both for short and long term outcomes and patients who have had this complication would be very keen for any intervention that may reduce the risk of this happening. It will eliminate a major source of risk for patients, improve quality of life, and produce immediate cost-savings for the NHS.

Compared to our current standard practice, which is limited as there is no direct visualisation of the bowel, the investigators feel this new technique will provide significantly more information to make an informed decision on an anastomosis and therefore lead to a reduction in leak rates. The current practice of an air-leak test is standard practice in the UK but a small number of centres have looked at endoscopic visualisation with less rigorous methodology (retrospective/non-randomised studies).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Undergoing colorectal resection involving the rectum
* Able to give informed consent to participate in trial
* American Society of Anesthesiologists (ASA) grade ≤ 3

Exclusion Criteria:

* Patients not undergoing colo-rectal/anal anastomosis e.g. abdominoperineal excision of rectum (APER), Hartmann's procedure.
* Patients undergoing synchronous colonic resections.
* Locally advanced rectal cancer requiring extended or multi-visceral excision.
* Recurrent rectal cancer
* Coexistent colorectal pathology e.g. synchronous cancers, inflammatory bowel disease.
* Previous pelvic radiotherapy for pathology unrelated to diagnosis with rectal cancer e.g. treatment for prostate cancer
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Clinical anastomotic leak | 60 days
  An anastomotic leak is defined as a defect of the intestinal wall at the anastomotic site leading to a communication between the intra- and extraluminal compartments. If there is clinical suspicion of an anastomotic leak (signs of peritonism on examination, rising inflammatory markers) a CT scan will be performed to confirm.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rossi, MBChB, Principal Investigator — University of Plymouth
Locations (1):
- University Hospitals Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No